CLINICAL TRIAL: NCT05852626
Title: Structuring Diabetes Care in Primary Health Care With Individualized Goals and Multidisciplinary Integration: A Cluster-randomized Clinical Trial for
Brief Title: Structuring of Diabetes Care in Primary Health Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20220197; 64538322.1.0000.5327 (Registry Identifier: Research ethics committee)
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Physicians

STUDY DESIGN:
Intervention Model Description: Cluster randomized clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Multimodal intervention in the primary care team that includes: redistribution of diabetes care between nurses and physicians, use of the individualized glycemic target calculator and implementation of minimum care recommendations
  Interventions: Other: Redistribution of diabetes care between nurses and physicians; Other: Individualized glycemic target; Other: Minimum care recomendations
- Control (Active Comparator): Usual follow-up in Primary Health Care (no intervention in the teams)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Redistribution of diabetes care between nurses and physicians — It will be proposed that nurses and physician share the clinical care of patients with type 2 diabetes, with complementing actions
  Arms: Intervention
Other: Individualized glycemic target — Define the target of individualized glycemic treatment for patients with the support of a tool on the website, which will encourage the intensification and de-intensification of treatment when appropriate
  Arms: Intervention
Other: Minimum care recomendations — It will be proposed to carry out the minimum necessary assessments that, annually, nurses and physicians must do to ensure the adequacy of quality indicators in the care of diabetes in the PHC
  Arms: Intervention
Other: No intervention — Primary care health teams will follow their rotine care of type 2 diabetes
  Arms: Control

SUMMARY:
The aim of this study is to evaluate the effectiveness of reorganization in Primary Health Care teams and individualized glycemic targets for type 2 diabetes.

DETAILED DESCRIPTION:
The prevalence of diabetes is increasing in parallel with the obesity epidemic. Diabetes is, therefore, a costly disease for individuals and healthcare system, generating expenses in its management and its complications. Also, it has significant social cost related to reduction of productivity. This study will evaluate the effectiveness of a multimodal intervention for Primary Health Care (PHC) teams to increase the nurse clinical role and implement individualized glycemic targets and care plan for type 2 diabetes through a pragmatic cluster-randomized clinical trial, with 1:1 allocation of health units in Porto Alegre, Brazil. Two study arms will be evaluated: 1) intervention group: will receive a set of proposed actions (redistribution of diabetes care between nurses and physicians, use of the individualized glycemic target calculator and implementation of care recommendations); 2) control group: usual follow-up in PHC.

ELIGIBILITY:
Health care unit:

Inclusion criteria

* Health unit has registered at least 50 users diagnosed with type 2 diabetes

Exclusion criteria:

* Health units that do not have a doctor and a nurse available on the same shift or do not have at least one doctor and a nurse willing to participate in the study.

Individuals:

Inclusion criteria

* Individuals with type 2 diabetes for at least one year
* In person diabetes consultation in the last six months

Exclusion criteria:

* Expected survival < one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who achieved individualized target HbA1c | 12 months
  Number of patients who achieved the individualized target HbA1c defined at baseline

SECONDARY OUTCOMES:
Percentage of clinical consultations carried out by nurses | 12 months
  Proportion of nursing consultations in relation to the total number of consultations (nurse and physician)
Foot evaluation | 12 months
  Total number of nursing consultations in which the feet were evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Schaan, Principal Investigator — UFRGS e HCPA
Locations (1):
- Ana Maria Frölich Matzenbacher, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
The data will be available from principal investigator upon reasonable request.